CLINICAL TRIAL: NCT01681940
Title: A Multi-Center, Open-Label Trial of the Long-term Efficacy and Safety of Lamazym for the Treatment of Patients With Alpha-Mannosidosis
Brief Title: Long-term Efficacy and Safety of Lamazym for the Treatment of Patients With Alpha-Mannosidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zymenex A/S (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rhLAMAN-04; 2011-004355-40 (EudraCT Number)
Record Dates: First submitted 2012-08-22; First posted 2012-09-10 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Alpha-Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamazym (Experimental): 1 mg/kg body weight
  Interventions: Drug: Lamazym

INTERVENTIONS:
Drug: Lamazym — ERT, i.v. infusions weekly
  Other Names: rhLAMAN; recombinant human alpha-mannosidase

SUMMARY:
The overall objective is to evaluate the long-term efficacy, safety and tolerability of repeated Lamazym i.v. treatment in patients 5-21 years of age with alpha-Mannosidosis

ELIGIBILITY:
Inclusion Criteria:

* The subject must have participated in the phase 1 trial (EudraCT number: 2010-022084-36) and phase 2a trial (EudraCT number: 2010-022085-26)
* Subject or subjects legally authorized guardian(s) must provide signed, informed consent prior to performing any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject)
* The subject and his/her guardian(s) must have the ability to comply with the protocol

Exclusion Criteria:

* The subject cannot walk without support
* Presence of known chromosomal abnormality and syndromes affecting psychomotor development, other than alpha-Mannosidosis
* History of bone marrow transplantation
* Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical conditions that, in the opinion of the Investigator, would preclude participation in the trial
* Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the trial.
* Pregnancy: Before the start of the treatment the investigators will decide whether or not there is a need for contraception. This assessment will be done through interviews with the patient and parents. The evaluation will be done continuously during the study
* Psychosis within the last 3 months
* Planned major surgery that, in the opinion of the investigator, would preclude participation in the trial
* Participation in other interventional trials testing IMP except for studies with Lamazym

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Reduction of Oligosaccharides in blood serum | 6 months
  Efficacy endpoint evaluation as change from baseline

SECONDARY OUTCOMES:
The number of steps climbed in 3 minutes (3-minute stair climb) | 6 months
  Efficacy endpoint evaluation as change from baseline
Reduction of Oligosaccharides in CSF | 6 months
  Efficacy endpoint evaluation as change from baseline
The distance walked in 6 minutes (6-minute walk test) | 6 months
  Efficacy endpoint evaluation as change from baseline
Pulmonary function | 6 months
  Efficacy endpoint evaluation as change from baseline
Adverse events | 1 week
  Safety endpoint assesed weekly throughout the trial
Development of clinically significant changes in vital signs and change in physical examination | 1 week
  Safety endpoint assesed weekly throughout the trial
Development of clinically significant changes in the clinical laboratory parameters (hematology, biochemistry and urinalysis) | 1 week
  Safety endpoint assesed weekly throughout the trial
Development of rhLAMAN antibodies and neutralizing/inhibitory antibodies | 1 week
  Safety endpoint assesed weekly throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Allan M Lund, MD, Principal Investigator — Copenhagen University Hospital, Center for Metabolic Diseases, Department for Clinical Genetics; Jens Fogh, Study Chair — Zymenex A/S
Locations (4):
- Kinderneurologie Metabole Ziekten, UZ Brussel, Laarbeeklaan 101, Brussels, Belgium
- Center for Metabolic Diseases, Department of Clinical Genetics, Juliane Marie Centre, Copenhagen University Hospital, Blegdamsvej 9, Copenhagen, Denmark
- Servicio de Pediatría, Hospital Materno Infantil, Reina Sofía, Avda Menéndez Pidal sn, Córdoba, Spain
- Genetic Medicine, 6th floor, St Mary's Hospital, Oxford Road,, Manchester, United Kingdom

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-004355-40